CLINICAL TRIAL: NCT07376915
Title: The Acute Effect of Graded Motor Imagery-Based Mental Preparation on Ankle Rehabilitation: A Pilot Clinical Study
Brief Title: Acute Effect of Graded Motor Imagery on Ankle Rehabilitation: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seda Ateş, physiotherapist, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/377
Record Dates: First submitted 2025-12-17; First posted 2026-01-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Ankle Instability; Healthy Controls

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- instability group (Experimental)
  Interventions: Other: graded motor imagery
- control group (Active Comparator)
  Interventions: Other: graded motor imagery

INTERVENTIONS:
Other: graded motor imagery — The Graded Motor Imagery (GMI) program will be applied six consecutive days nd will consist of three progressive stages:
  Laterality Training:
  Participants will perform right-left ankle discrimination tasks using validated foot and ankle images. Accuracy and response time will be recorded.
  Motor Imagery:
  Participants will mentally rehearse ankle movements such as dorsiflexion, plantarflexion, inversion, and eversion without performing the motion. Imagery tasks will progress from simple movements to functional patterns based on tolerance.
  Mirror Therapy:
  A mirror will be placed in the midsagittal plane, allowing participants to view the reflection of the non-affected ankle while performing movements. The visual illusion of normal movement is intended to improve motor control and proprioception.

SUMMARY:
The primary aim of this study is to evaluate the immediate and short-term effects of the Graded Motor Imagery (GMI) method on individuals with chronic ankle instability (CAI). In this context, the effects of the Graded Motor Imagery intervention on pain level, muscle stiffness, muscle strength, functional performance, and subjective instability level will be investigated. Additionally, these effects will be comparatively analyzed with an age- and sex-matched control group consisting of healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years.
* Diagnosed with chronic ankle instability (CAIT ≤ 24).
* History of an acute ankle sprain occurring more than 3 months prior to enrollment.
* Has not received ankle rehabilitation treatment.
* Voluntarily participated in this study

Exclusion Criteria:

* Vestibular or neurological disorders
* Other lower extremity injuries
* History of surgery

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02-09 (Actual); Primary Completion 2026-06-09 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
Subjective Instability (CAIT) | baseline
  A valid-reliable questionnaire that questions the perceived instability in daily life and sports activities.
  Clinical Significance: ≥ 3 point increase is considered clinically significant
Subjective Instability (CAIT) | 1-week post-intervention
  A valid-reliable questionnaire that questions the perceived instability in daily life and sports activities.
  Clinical Significance: ≥ 3 point increase is considered clinically significant
Ground Reaction Force & Static Balance (ForceDecks) | baseline
  Device: ForceDecks dual force platform.
  1. Single-Leg Jump Test* Values: Net vertical ground reaction force (N·kg-¹), flight time (ms), asymmetry (%).
  2. Single-Leg Static Balance* Values: Total sway path (mm), ellipse area (mm²).
  Clinical Importance:* Captures short-term changes in neuromuscular control and explosive strength in a detailed manner.
Ground Reaction Force & Static Balance (ForceDecks) | 1-week post-intervention
  Device: ForceDecks dual force platform.
  1. Single-Leg Jump Test* Values: Net vertical ground reaction force (N·kg-¹), flight time (ms), asymmetry (%).
  2. Single-Leg Static Balance* Values: Total sway path (mm), ellipse area (mm²).
  Clinical Importance:* Captures short-term changes in neuromuscular control and explosive strength in a detailed manner.

SECONDARY OUTCOMES:
Muscle Stiffness (Myoton PRO) | baseline
  Tonic stiffness (N·m-¹) reflects the passive mechanical properties of muscle tissue. The device applies a 0.4 N mechanical impulse to the skin and records the resulting tissue oscillation response. In this study, data will be recorded as the average of 3 impulses.
  Clinical Importance: Acute changes in stiffness are considered an indirect indicator of neuroplastic responses in proprioception and motor control.
Muscle Stiffness (Myoton PRO) | 1-week post-intervention
  Tonic stiffness (N·m-¹) reflects the passive mechanical properties of muscle tissue. The device applies a 0.4 N mechanical impulse to the skin and records the resulting tissue oscillation response. In this study, data will be recorded as the average of 3 impulses.
  Clinical Importance: Acute changes in stiffness are considered an indirect indicator of neuroplastic responses in proprioception and motor control.
Muscle Strength Assessment - Isokinetic dynamometer (Isoforce) | baseline
  Parameter: Concentric inversion-eversion peak torque (Nm) at 60°·s-¹ Objectively measures agonist-antagonist muscle performance around the ankle joint.
  Clinical Significance:* Improvements in strength contribute to functional stability and a reduced risk of re-injury.
Muscle Strength Assessment - Isokinetic dynamometer (Isoforce) | 1-week post-intervention
  Parameter: Concentric inversion-eversion peak torque (Nm) at 60°·s-¹ Objectively measures agonist-antagonist muscle performance around the ankle joint.
  Clinical Significance:* Improvements in strength contribute to functional stability and a reduced risk of re-injury.
Pain Level | baseline
  Visual Analog Scale (VAS, 0-10 cm): 0 = "no pain," 10 = "unbearable pain"; the participant marks the scale before and after the session.
Pain Level | 1-week post-intervention
  Visual Analog Scale (VAS, 0-10 cm): 0 = "no pain," 10 = "unbearable pain"; the participant marks the scale before and after the session.
Functional Performance | baseline
  Star Excursion Balance Test (SEBT) Parameter: Normalized reach distance in three primary directions (anteromedial, medial, posteromedial), expressed as a percentage of leg length.
  Clinical Significance: Assesses dynamic balance and lateral load-transfer capacity; asymmetries in individuals with chronic ankle instability (CAI) may serve as prognostic indicators.
Functional Performance | 1-week post-intervention
  Star Excursion Balance Test (SEBT) Parameter: Normalized reach distance in three primary directions (anteromedial, medial, posteromedial), expressed as a percentage of leg length.
  Clinical Significance: Assesses dynamic balance and lateral load-transfer capacity; asymmetries in individuals with chronic ankle instability (CAI) may serve as prognostic indicators.

CONTACTS AND LOCATIONS:
Overall Officials: SEZEN KARABÖRKLÜ ARGUT, Assistant Professor, PhD, Study Director — Istanbul University-Cerrahpaşa, Faculty of Health Sciences
Locations (1):
- İstanbul Üniversitesi-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim KM, Estepa-Galego A, Estudilo-Martínez MD, Castelote-Cabalero Y, Cruz-Díaz D. Comparative Effects of Neuromuscular- and Strength-Training Protocols on Pathomechanical, Sensory-Perceptual, and Motor-Behavioral Impairments in Patients with Chronic Ankle Instability: Randomized Contro led Trial. Healthcare (Basel). 2022 Jul 22;10(8):1364. doi: 10.3390/healthcare10081364. PMID: 35893186; PMCID: PMC9394255.
- [Background] Naderi A, Ahi K. Comparative analysis of land-based vs. water-based balance training on quality of life and physical and psychological deficits in athletes with chronic ankle instability: a randomized contro led trial. BMC Sports Sci Med Rehabil. 2025 Jan 20;17(1):9. doi: 10.1186/s13102-024-01049-3. PMID: 39828772; PMCID: PMC11744859.
- [Background] David P, Halimi M, Mora I, Doutrelot PL, Petitjean M. Isokinetic testing of evertor and invertor muscles in patients with chronic ankle instability. J Appl Biomech. 2013 Dec;29(6):696-704. doi: 10.1123/jab.29.6.696. Epub 2013 Jan 18. PMID: 23343782.
- [Background] Wright CJ, Linens SW, Cain MS. Establishing the Minimal Clinical Important Difference and Minimal Detectable Change for the Cumberland Ankle Instability Tool. Arch Phys Med Rehabil. 2017 Sep;98(9):1806-1811. doi: 10.1016/j.apmr.2017.01.003.
- [Background] Moseley GL. Graded motor imagery for pathologic pain: a randomized controled trial. Neurology. 2006 Dec 26;67(12):2129 34. doi: 10.1212/01.wnl.0000249112.56935.32. Epub 2006 Nov 2. PMID: 17082465.